CLINICAL TRIAL: NCT02566837
Title: Ultrasound Guidance to Alleviate the Pain Associated With Intramuscular Injections of Botulinum Toxin in Spastic Patients
Brief Title: Use of Ultrasound in Injections of Botulinum Toxin
Acronym: TOXINECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11 425 03; 2012-A00004-39 (Registry Identifier: Agence National du Médicament et des Produits de santé)
Record Dates: First submitted 2015-08-18; First posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Spasticity
Keywords: ultrasound; Electrical stimulation guidance; botulinum toxin
MeSH Terms: conditions — Muscle Spasticity | interventions — High-Energy Shock Waves; Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ELEC (Active Comparator): electrical stimulation guidance
  Interventions: Procedure: electrical stimulation
- ECHO (Experimental): ultrasound guidance
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — ultrasound imaging to guide the intramuscular injections of botulinum toxin : Ultrasound is used to identify the target muscle, and for guiding the insertion of the needle in the muscle. Once the needle is positioned, the botulinum toxin is injected
  Arms: ECHO
Procedure: electrical stimulation — electrical stimulation (reference technique currently recommended over muscle palpation and anatomical landmarks) to guide intramuscular injections of botulinum toxin. Intramuscular injection is carried out in register with the zone where is located the theoretically target muscle. Electrical stimulation (mediated by the tip of the needle) used to verify the correct position of the needle, and reposition it if necessary. Once the needle is correctly positioned, the botulinum toxin is injected.
  Arms: ELEC

SUMMARY:
Intramuscular injections of botulinum toxin are currently the best focal treatment of spasticity, with clearly defined indications and role. French and European recommendations focus on the toxin's mode of administration, which must be as precise as possible. The toxin's specific action on motor endplates (blocking the release of acetylcholine) shows the importance of targeted injections within the muscle belly. The pain caused by these injections is due partly the number of injections (up to 30 in a single session), and partly to the use of electrical stimulation guidance. Prevention and alleviation of the pain caused by these injections have become a regulatory obligation since the law of 4 March 2002 relating to the rights of patients and the quality of the health system (" Any person has the right to receive relief from pain, which must, under all circumstances, be prevented, evaluated, taken into account and treated … ").

DETAILED DESCRIPTION:
Electrical stimulation guidance is generally used nowadays, and is recommended over the use of palpation and anatomical landmarks. However, electrical stimulation has its limits. It is sometimes poorly tolerated by patients as it causes pain, which is greater in muscles less responsive to such stimulation and requiring a stronger electrical current. The pain also increases with the number of injections performed in a single session. Electrical stimulation does not guarantee for certain that the needle is placed within the muscle, as a stimulation of the aponeurosis may cause the muscle to contract through the excitation of motor branches entering the muscle. The injection of botulinum toxin in the aponeurosis does not provide a satisfactory effect and may render the injection ineffective. In some patients, the muscle to inject may present some degree of retraction with fat degeneration, which reduces its sensitivity to electrical stimulation. Individual patients may also respond poorly or not at all to electrical stimulation, which causes technical and treatment problems. Finally, certain muscles are difficult to locate by electrical stimulation because their contraction produces only weak mechanical effects (e.g. short muscles such as the interossei muscles). All these factors explain why ultrasound imaging provides an interesting alternative guidance technique for botulinum toxin injections. In most cases, it can replace electrical stimulation altogether, and thus avoid the pain it causes. Ultrasound guidance is already recommended in pediatric patients to improve their comfort during the injections. In our study, the patient's comfort during the injection was chosen as the main endpoint because it has already been demonstrated in children and because the investigators feel it is an essential aspect of our routine practice. Moreover, ultrasound imaging helps locate accurately the muscle to be injected. Once the tip of the needle has been located, it can be tracked during the injection, and guided to the muscle belly. Previous studies have already shown that this technique improves the efficacy of the injections. Ultrasound imaging is also interesting when the muscles to be injected are located in a deep plane or close to vital structures, such as nerves, arteries, or veins (e.g. piriformis or psoas). All these considerations have been studied in children and should be validated in adult spastic patients as well.

Therefore, the investigators will compare ultrasound guidance to electrical stimulation guidance in routine clinical practice. This study will be carried out in adult spastic patients who may receive botulinum toxin injections in the Service of Physical Medicine and Rehabilitation of University Teaching Hospital. The aim is to analyse the advantages of this injection technique under current practice conditions.

The evaluating physician (blinded) will conduct a clinical examination of the patients before the injections, and 6 to 8 weeks after the injection of botulinum toxin. The pain associated with the toxin injections will be evaluated after the injections and during the follow-up visit, using the vertical indexed VAS and the Face Pain Scale. The spasticity will be evaluated on the Tardieu scale before the injections and during the follow-up visit. The duration of the botulinum toxin injections will be measured. Finally, functional objectives will be determined prior to the injections. The GAS (Goal Attainment Scaling) methodology will be used during the follow-up visit to determine whether these objectives have been met or not.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patient with a spasticity associated with a central neurological lesion caused by vascular hemiplegia, head trauma, sequelae of cerebral anoxia, multiple sclerosis, spinal cord injury, or cerebral palsy.
* Patient with a spasticity with an indication for a focal treatment with intramuscular injections of botulinum toxin, and associated with:
* Functional discomfort
* Tardieu score ≥1 for one or several muscles in the upper and/or lower limbs
* Patient naive to intramuscular botulinum toxin injections, and in whom the physician wishes to use the Speywood botulinum toxin (Dysport).
* Patient able to self-evaluate the pain on a VAS and understand three successive instructions, such as those used in the Mini Mental Status(MMS).
* Patient able to give his/her consent to participate.
* Patients able to provide a signed informed consent freely for the study protocol and data collection.
* Patient with a recognised Long-Term Illness, and thus necessarily covered by the social security.

EXCLUSION CRITERIA:

* General contra-indications of botulinum toxin:

  * History of myasthenia or Lambert-Eaton syndrome
  * History of neuromuscular disease
  * Previous surgery with curarization less than a month ago
  * Treatment with aminosides, aminoquinoleines or cyclosporine
* Progressive neurological disease at the time of inclusion
* Anticoagulant treatment: heparin administered with an electrical syringe or anticoagulant therapy with effective doses
* Legal incompetence (judicial protection, guardianship)
* Subject participating in another study, with an exclusion period on-going at the time of the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
pain caused by the injections | inclusion
  pain evaluated by vertical visual analogue scale indexed

SECONDARY OUTCOMES:
Compare the pain felt by the patient | 7 weeks after inclusion
  pain evaluated by vertical visual analogue scale indexed
Compare the pain felt by the patient | 7 weeks after inclusion
  pain evaluated by the Face Pain Scale
reduction of spasticity | 6-8 weeks after inclusion
  using Tardieu scale
Compare the time required to perform the injections of botulinum toxin under ultrasound guidance and under electrical guidance. | inclusion
  Time to perform the injections will be notified in minutes
Compare the efficacy of the injections of botulinum toxin in terms of functional gain. | 6-8 weeks after inclusion
  efficacy was evaluated by Goal Attainment Scaling (GAS)

CONTACTS AND LOCATIONS:
Overall Officials: David GASQ, MD, Principal Investigator — Service d'explorations fonctionnelles - Hôpital Rangueil
Locations (1):
- Rangueil Hospital, Toulouse, France